CLINICAL TRIAL: NCT01159756
Title: To Assess the Safety and Efficacy of Travacom in Patients With Uncontrolled Intraocular Pressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-10-01
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-01

CONDITIONS: Uncontrolled Intraocular Pressure
Keywords: Travacom; Glaucoma; Travoprost; Timolol
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Travacom (Experimental): Travacom ophthalmic solution
  Interventions: Drug: Travacom

INTERVENTIONS:
Drug: Travacom — Travacom ophthalmic solution (1 drop per day)

SUMMARY:
This study is a multi-site, unmasked phase IV study. Travacom(R) is a combination topical ocular agent, containing travoprost and timolol, which lower intraocular pressure (IOP) by complementary mechanisms of action. The safety and efficacy of both travoprost and timolol have been established as single and adjunctive therapy in well-controlled clinical studies in thousands of patients diagnosed with open angle glaucoma (OAG) or ocular hypertension. The objective of this study is to assess the safety and efficacy of changing to Travacom from prior pharmacotherapy in uncontrolled patients with open-angled glaucoma or ocular hypertension across India.

ELIGIBILITY:
Inclusion Criteria:

* Must have a clinical diagnosis of ocular hypertension, primary open-angle or pigment dispersion glaucoma in both eyes.
* Must be willing to discontinue the use of all other ocular hypotensive medications prior to receiving the study medication for the entire course of the study.
* Must be able to follow instructions and be willing and able to attend all study visits.

Exclusion Criteria:

* A known medical history of allergy, hypersensitivity or poor tolerance to any component of Travacom that is deemed clinically significant in the opinion of the Principle Investigator.
* Any abnormality preventing reliable applanation tonometer in either eye. Corneal dystrophies.
* Any opacity or subject uncooperativeness that restricts adequate examination of the ocular fundus or anterior chamber of either eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2010-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Primary efficacy: Change in IOP at the final visit from prior beta-blocker monotherapy (Timolol 0.5% only) | Baseline to Visit 3 (Week 6-8)
  To assess the efficacy of changing to Travacom from prior pharmacotherapy in uncontrolled patients with open-angled glaucoma or ocular hypertension.
Safety: Adverse Events. | Baseline to Visit 3 (Week 6-8)
  To assess the safety of changing to Travacom from prior pharmacotherapy in uncontrolled patients with open-angled glaucoma or ocular hypertension.
Secondary efficacy: Percentage of subjects at target IOP (</ 18 mmHg), regardless of prior therapy. | Baseline to Visit 3 (Week 6-8)
  To assess the efficacy of changing to Travacom from prior pharmacotherapy in uncontrolled patients with open-angled glaucoma or ocular hypertension.

CONTACTS AND LOCATIONS:
Locations (1):
- Disha Eye Hospitals, Kolkata, India